CLINICAL TRIAL: NCT00061568
Title: Nonmyeloablative Allogeneic Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Severe Congenital Anemias Including Sickle Cell Disease (SCD) and B-Thalassemia
Brief Title: Improving the Results of Bone Marrow Transplantation for Patients With Severe Congenital Anemias
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030170; 03-H-0170
Record Dates: First submitted 2003-05-29; First posted 2003-05-29 (Estimated); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Congenital Hemolytic Anemia; Sickle Cell Disease
Keywords: Stem Cell Transplant; Low Dose Radiation; Alemtuzumab (Campath); Sirolimus (Rapamune); Donor Apheresis; Sickle Cell Anemia (SCA); Beta-Thalassemia
MeSH Terms: conditions — Anemia, Hemolytic, Congenital; Anemia, Sickle Cell; beta-Thalassemia | interventions — Transplantation; Alemtuzumab; Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants (Experimental): Nonmyeloablative transplant regiment, consisting of alemtuzumab (1 mg/kg in divided doses), total-body irradiation (300 cGy), sirolimus, and infusion of unmanipulated filgrastim mobilized peripheral blood stem cells from human leukocyte antigen-matched siblings.
  Interventions: Procedure: Peripheral blood hematopoietic progenitor cell (PBPC) transplant; Drug: Alemtuzumab; Drug: Sirolimus
- Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor (Experimental): Participants received Filgrastim to mobilize peripheral blood stem cells for apheresis collection. Collected stem cells of donor will then be infused to HLA matched sibling.
  Interventions: Procedure: Peripheral blood hematopoietic progenitor cell Apheresis

INTERVENTIONS:
Procedure: Peripheral blood hematopoietic progenitor cell (PBPC) transplant — Peripheral blood hematopoietic progenitor cell (PBPC) transplant
  Arms: Participants with Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Drug: Alemtuzumab — Alemtuzumab
  Other Names: Campath
  Arms: Participants with Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Procedure: Peripheral blood hematopoietic progenitor cell Apheresis — Donor-Peripheral blood hematopoietic progenitor cell (PBPC) apheresis
  Arms: Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor
Drug: Sirolimus — Sirolimus
  Other Names: Rapamune
  Arms: Participants with Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants

SUMMARY:
People with severe congenital anemias, such as sickle cell anemia and beta-thalassemia, have been cured with bone marrow transplantation (BMT). The procedure, however, is limited to children younger than the age of 16 because the risks are lower for children than for adults.

The purpose of this study is to explore the use of a BMT regimen that, instead of chemotherapy, uses a low dose of radiation, combined with two immunosuppressive drugs. This type BMT procedure is described as nonmyeloablative, meaning that it does not destroy the patient s bone marrow. It is hoped that this type of BMT will be safe for patients normally excluded from the procedure because of their age and other reasons.

To participate in this study, patients must be between the ages of 18 and 65 and have a sibling who is a well-matched stem-cell donor. Beyond the standard BMT protocol, study participants will undergo additional procedures. The donor will receive G-CSF by injection for five days; then his or her stem cells will be collected and frozen one month prior to BMT. Approximately one month later, the patient will be given two immune-suppressing drugs, Campath 1-H and Sirolimus, as well as a single low dose of total body irradiation and then the cells from the donor will be infused.

Prior to their participation in this study, patients will undergo the following evaluations: a physical exam, blood work, breathing tests, heart-function tests, chest and sinus x-rays, and bone-marrow sampling.

...

DETAILED DESCRIPTION:
Nonmyeloablative allogeneic peripheral blood stem cell (PBSC) transplants are currently being investigated in phase I/II trials assessing engraftment, efficacy, and toxicity at a number of transplant centers. Preliminary data have shown a high rate of complete donor engraftment with a relatively low toxicity profile. The decreased risk of transplant-related complications associated with nonmyeloablative transplants expands eligibility to patients with nonmalignant hematological disorders curable by allogeneic transplantation; however, significant toxicity with current regimens persists including severe graft versus host disease (GVHD) leading to significant morbidity and mortality. Moreover, mixed chimerism has been shown to be sufficient to induce clinical remissions in children with nonmalignant hematologic disorders undergoing conventional allogeneic transplantation. Therefore, newer regimens need to be developed that are more applicable to patients with non-malignant disorders in whom no graft vs. leukemia effect is needed, and where mixed chimerism is sufficient for disease amelioration.

In this protocol, we propose transplantation in patients with severe beta-globin disorders including sickle cell disease (SCD), and beta-thalassemia, considered at high risk for complications from or ineligible for standard BMT, with allogeneic PBSCs from an HLA identical sibling using a novel immunosuppressive regimen without myeloablation in an attempt to further decrease the transplant related morbidity/mortality. The low intensity nonmyeloablative conditioning regimen will consist of low dose radiation, Alemtuzumab (Campath) and Sirolimus (Rapamune) as a strategy to provide adequate immunosuppression to allow sufficient engraftment for clinical remission with a lower risk of GVHD development. T-cell replete, donor-derived, granulocyte colony stimulating factor (filgrastim, G-CSF) mobilized PBSCs will be used to establish hematopoietic and lymphoid reconstitution.

The primary endpoint of this study is treatment success at one year, defined as full donor type hemoglobin on hemoglobin electrophoresis for patients with SCD and transfusion-independence for patients with beta-thalassemia. Other end points include degree of donor-host chimerism necessary for long-term graft survival and disease amelioration, incidence of acute and chronic graft-vs-host disease (GVHD), incidence of graft rejection, transplant related morbidity, as well as disease-free and overall survival.

ELIGIBILITY:
* INCLUSION CRITERIA:

RECIPIENTS:

Must fulfill one disease category from below:

DISEASE SPECIFIC:

Patients with sickle cell disease at high risk for disease related morbidity or mortality, defined by having irreversible end organ damage (A, B, C, D or E) or potentially reversible complication(s) not ameliorated by hydroxyurea (F):

A. Stroke defined as a clinically significant neurologic event that is accompanied by and infarct on cerebral MRI

OR

an abnormal trans-cranial Doppler examination ( greater than or equal to 200m/s);

OR

B. Sickle cell related renal insufficiency defined by a creatinine level greater than or equal to 1.5 times the upper limit of normal and kidney biopsy consistent with sickle cell nephropathy OR nephritic syndrome OR creatinine clearance less than 60mL/min/1.73m(2) for patients less than or equal to 16 years of age or less than 50mL/min for patients greater than or equal to 16 years of age OR requiring peritoneal or hemodialysis

OR

Age is less than or equal to 5 years of age with the upper limit of normal serum creatinine 0.8mg/dl

Age is greater than 5 years or less than or equal to 10 years of age with the upper limit of normal serum creatinine 1.0mg/dl

Age is greater than 10 years and less than or equal to 15 years of age the the upper limit of normal serum creatinine 1.2mg/dl

Age greater than 15 years of age with the upper limit of normal serum creatinine 1.3mg/dl

C. Tricuspid regurgitant jet velocity (TRV) of greater than or equal to 2.5m/s in patients greater than or equal to 18 years of age at least 3 weeks after a vaso-occlusive crisis, OR

D. Recurrent tricorporal priapism defined as at least two episodes of an erection lasting greater than or equal to 4 hours involving the corpora cavernosa and corpus spongiosa, OR

E. Sickle hepatopathy defined as EITHER ferritin greater than 100mcg/L OR direct bilirubin greater than 0.4 mg/dL at baseline in patients greater than or equal to 18 years of age; OR

F. Any one of the below complications:

1. Vaso-occlusive crisis:

   * Eligible for hydroxyurea; at least 3 hospital admissions in the last year
   * Eligible for HSCT; More than 1 hospital admission per year while on therapeutic dose of hydroxyurea
2. Acute Chest Syndrome (ACS):

   * Eligible for hydroxyurea: 2 prior ACS while greater than 3 years of age and adequately treated for asthma
   * Eligible for HSCT: any ACS while on hydroxyurea*
3. Osteonecrosis of 2 or more joints:

   * Eligible for hydroxyurea: And significantly affecting their quality of life by Karnofsky score 50-60
   * Eligible for HSCT: And on hydroxyurea* where total hemoglobin increase less than 1g/dL or fetal hemoglobin increases less than 2.5 time the baseline level
4. Red cell alloimmunization:

   * Eligible for hydroxyurea: Transfusion dependent
   * Eligible for HSCT: Total hemoglobin increase less than 1 g/dL while on hydroxyurea*

     * hydroxyurea at therapeutic dose

   Patients with beta-thalassemia who have grade 2 or 3 iron overload, determined by the presence of 2 or more of the following:
   * portal fibrosis by liver biopsy
   * inadequate chelation history (defined as failure to maintain adequate compliance with chelation with desferoxamine initiated within 18 months of the first transfusion and administered subcutaneously for 8-10 hours at least 5 days each week)
   * Hepatomegaly of greater than 2 cm below the costochondral margin

   NON-DISEASE SPECIFIC:
   * Ages greater than or equal to 4 years
   * 6/6 HLA matched family donor available
   * Ability to comprehend and willing to sign an informed consent, assent obtained from minors
   * Negative serum beta-HCG
   * Pediatric patients less than 16 years of age must decline myeloablative bone marrow transplantation

   DONOR:

   Donor deemed suitable and eligible, and willing to donate per clinical evaluations, who are additionally willing to donate blood for research and undergo a neuropsychological test. Donors will be evaluated in accordance with existing Standard NIH Policies and Procedures for determination of eligibility and suitability for clinical donation under a separate NHLBI protocol. Note that participation in this study is offered to all donors, but is not required for a donor to make a stem cell donation, so it is possible that not all donors will enroll onto this study.

   EXCLUSION CRITERIA:

   RECIPIENT:

   (Any of the following would exclude the subject from participating)

   ECOG performance status of 3 or more or Lansky performance status of less than 40.

   Diffusion capacity of carbon monoxide (DLCO) less than 35% predicted. (corrected for hemoglobin and alveolar volume)

   Baseline oxygen saturation or less than 85 % or PaOa2 less than 70

   Left ventricular ejection fraction: less than 35% estimated by ECHO.

   Transaminases greater than 5 times the upper limit of normal for age

   Evidence of uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen

   Major anticipated illness or organ failure incompatible with survival from PBSC transplant.

   Pregnant or lactating

   Major ABO mismatch

   DONOR:

   None

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-07-16 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol is available to be shared upon request to PI.
Supporting Information: Study Protocol
Time Frame: Immediately
Access Criteria: Protocol is available to be shared upon request to PI.

REFERENCES:
- [Background] Wayne AS, Schoenike SE, Pegelow CH. Financial analysis of chronic transfusion for stroke prevention in sickle cell disease. Blood. 2000 Oct 1;96(7):2369-72. PMID 11001885
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Charache S, Terrin ML, Moore RD, Dover GJ, Barton FB, Eckert SV, McMahon RP, Bonds DR. Effect of hydroxyurea on the frequency of painful crises in sickle cell anemia. Investigators of the Multicenter Study of Hydroxyurea in Sickle Cell Anemia. N Engl J Med. 1995 May 18;332(20):1317-22. doi: 10.1056/NEJM199505183322001. PMID 7715639
- [Derived] Inam Z, Jeffries N, Link M, Coles W, Pollack P, Luckett C, Phang O, Harvey E, Martin T, Farrey T, Tisdale JF, Hsieh MM. Two Nonmyeloablative HLA-Matched Related Donor Allogeneic Hematopoietic Cell Transplantation Regimens in Patients with Severe Sickle Cell Disease. Transplant Cell Ther. 2025 May;31(5):305-318. doi: 10.1016/j.jtct.2025.02.021. Epub 2025 Feb 24. PMID 40010689
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296
- [Derived] Hsieh MM, Fitzhugh CD, Weitzel RP, Link ME, Coles WA, Zhao X, Rodgers GP, Powell JD, Tisdale JF. Nonmyeloablative HLA-matched sibling allogeneic hematopoietic stem cell transplantation for severe sickle cell phenotype. JAMA. 2014 Jul 2;312(1):48-56. doi: 10.1001/jama.2014.7192. PMID 25058217
- [Derived] Hsieh MM, Kang EM, Fitzhugh CD, Link MB, Bolan CD, Kurlander R, Childs RW, Rodgers GP, Powell JD, Tisdale JF. Allogeneic hematopoietic stem-cell transplantation for sickle cell disease. N Engl J Med. 2009 Dec 10;361(24):2309-17. doi: 10.1056/NEJMoa0904971. PMID 20007560
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-H-0170.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor: Participants received filgrastim to mobilize peripheral blood stem cells for apheresis collection. Collected stem cells of donor will then be infused to HLA matched recipient of stem cell transplant.
Period: Overall Study
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor
Started | 62 | 68
Completed | 43 | 68
Not Completed | 19 | 0
Not completed — Lost to Follow-up | 12 | 0
Not completed — Death | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor | Total
Number analyzed (Participants) | 62 | 68 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 12 | 16
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 51
  Male | 41 | 38 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 56 | 61 | 117
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 58 | 110
  White | 4 | 4 | 8
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 62 | 68 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience Treatment Success Following Stem Cell Transplant
Description: Number of participants that experience treatment success at one year following stem cell transplant. Treatment success is defined as full donor type hemoglobin on hemoglobin electrophoresis for patients with sickle cell disease and transfusion-independence for patients with beta-thalassemia.
Time Frame: Up to 1 year
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Participants with Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants | 53

2. Secondary Outcome: Mean Myeloid Chimerism Level
Description: Mean Myeloid Chimerism Level in participants following stem cell transplant.
Time Frame: up to 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % of Donor Chimerism
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
% of Donor Chimerism
  Myeloid Chimerism | 90.1 (2.8)
  CD3+ Chimerism | 55.0 (3.5)

3. Secondary Outcome: Number of Participants Who Developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as Defined by CIMBTR Criteria for Organ Stages of Acute GVHD.
Description: Number of participants who developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grades are defined as:
  Grade I: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants
  Grade I Acute Graft Verses Host Disease | 0
  Grade II Acute Graft Verses Host Disease | 0
  Grade III Acute Graft Verses Host Disease | 0
  Grade IV Acute Graft Verses Host Disease | 0

4. Secondary Outcome: Number of Participants Who Developed Limited or Extensive Chronic GVHD
Description: Number of participants who developed Limited or Extensive Chronic Graft vs Host Disease (GVHD).
  Limited disease is characterized by localized skin involvement and/or evidence of hepatic dysfunction. Limited disease is associated with a favorable outcome without systemic therapy, while extensive disease patients have an unfavorable outcome.
  Extensive chronic GVHD is defined as GVHD occurring after day 100 that did not meet the definition of limited chronic GVHD. Extensive disease presents either with generalized skin involvement, or with localized skin involvement or hepatic dysfunction plus at least one of the following:
  Liver histology showing chronic progressive hepatitis, bridging necrosis, or cirrhosis Involvement of the eye (Schirmer's test with less than 5 mm wetting) (see "Diagnosis and classification of Sjögren's syndrome") Involvement of minor salivary glands or oral mucosa (as demonstrated on labial or mucosal biopsy specimen) Involvement of any other target organ
Time Frame: Day 100 up to 3 Years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants
  Limited Chronic Graft vs Host Disease | 0
  Extensive Chronic Graft vs Host Disease | 0

5. Secondary Outcome: Number of Participants With Regimen Failure
Description: Number of participants with regimen failure. Regimen failure is defined as those participants that experienced graft verses host disease or relapse of sickle cell disease or beta-thalassemia.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants | 9

6. Secondary Outcome: Number of Participants With Disease-free Survival
Description: Number of participants with disease-free survival, as defined by: alive and free of acute complications related to sickle cell disease or beta-thalassemia.
Time Frame: Up to 2 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants | 51

7. Secondary Outcome: Number of Participants Overall Survival
Description: Number of participants overall survival at year 1 and year 2. Overall survival is defined as participants alive at 1 and 2 years following stem cell transplant.
Time Frame: 1 year and 2 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants
  Participants alive at 1 year post stem cell transplant | 61
  Participants alive at 2 years post stem cell transplant | 61

8. Secondary Outcome: Number of Participants That Experienced a Transplant-related Mortality
Description: Number of participants that experienced a transplant related mortality, as defined as death from causes other than relapse (such as: GVHD, toxicity, infection, other and unknown causes).
Time Frame: Up to 2 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants
Number analyzed (Participants) | 62
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor
All-Cause Mortality (participants affected / at risk) | 6/62 | 0/68
Serious Adverse Events (participants affected / at risk) | 44/62 | 6/68
Other Adverse Events (participants affected / at risk) | 13/62 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants (N=62) | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor (N=68)
Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Relapse of sickle cell disease (Congenital, familial and genetic disorders) | 6 (6) | 0 (0)
Babesiosis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (8) | 0 (0)
Sirolimus associated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Sirolimus related arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Clostridioides difficile colitis (Infections and infestations) | 1 (2) | 0 (0)
Sirolimus associated fever (General disorders) | 1 (1) | 0 (0)
Pancreatitis (Infections and infestations) | 1 (1) | 0 (0)
Abscess versus infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Thromboembolism (Vascular disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Reticulocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Narcotic dependence (General disorders) | 3 (6) | 0 (0)
Strangulated ventral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dialysis catheter thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal bleed on warfarin (Gastrointestinal disorders) | 1 (1) | 0 (0)
Herpes simplex virus (Infections and infestations) | 1 (1) | 0 (0)
Temporary left sided weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypotension post transfusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Right forearm compartment syndrome (Vascular disorders) | 1 (1) | 0 (0)
Cytomegalovirus reactivation (Infections and infestations) | 1 (1) | 0 (0)
Anti-D hemolysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Intracranial Bleed from Moya-Moya disease (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary complication of unknown etiology (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Factor 8 inhibitor (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Intracranial Bleed (Vascular disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever with unclear etiology (General disorders) | 2 (2) | 0 (0)
Apthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 0 (0)
Vaso-occlusive pain crisis (Congenital, familial and genetic disorders) | 2 (3) | 0 (0)
Pain post bone marrow harvest (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Acute psychotic episode (Psychiatric disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 3 (3) | 0 (0)
Liver biopsy (Surgical and medical procedures) | 2 (2) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Acute Graft Verses Host Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (2) | 0 (0)
Chronic myelogenous leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prosthetic and surrounding tissue bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary thromboendarterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Non Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hip replacement (Surgical and medical procedures) | 1 (2) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Right shoulder replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Prolonged bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Citrate toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arterio-venous fistula from line placement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis Secondary to Salmonella Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Severe Beta-globin Disorders in Allogeneic Peripheral Blood Stem Cell Transplants (N=62) | Human Leukocyte Antigens (HLA) Matched Related Stem Cell Donor (N=68)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Weight gain (Investigations) | 5 (5) | 0 (0)
Hypothyroid (Endocrine disorders) | 3 (3) | 0 (0)
Hyperthyroid (Endocrine disorders) | 3 (3) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 13 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT00061568/Prot_SAP_000.pdf